CLINICAL TRIAL: NCT00606086
Title: A Phase 2 Randomized, Open Label, Multi-center, Therapeutic Trial of the Efficacy, Immunogenicity, and Safety of GI-5005; an Inactivated Recombinant Saccharomyces Cerevisiae Expressing a Hepatitis C Virus NS3-Core Fusion Protein, Combined With Pegylated Interferon Plus Ribavirin Standard of Care Therapy Versus Standard of Care Alone, and GI-5005 Salvage of Standard of Care Failures, in Patients With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Safety and Efficacy of the Therapeutic Vaccine GI-5005 Combined With Pegylated Interferon Plus Ribavirin Standard of Care Therapy Versus Standard of Care Alone in Patients With Genotype 1 Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlobeImmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI-5005-02
Record Dates: First submitted 2008-01-18; First posted 2008-02-01 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Genotype 1 Chronic Hepatitis C
Keywords: Hepatitis, HCV, Liver disease, HepC
MeSH Terms: conditions — Hepatitis; Hepatitis C; Liver Diseases | interventions — GI 5005; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): GI-5005 monotherapy continuing on to triple therapy
  Interventions: Drug: GI-5005
- 2 (Active Comparator): Standard of care alone
  Interventions: Drug: GI-5005; Drug: Pegylated Interferon and Ribavirin

INTERVENTIONS:
Drug: GI-5005 — 40YU, subcutaneous
  Other Names: Pegasys and Ribavirin
Drug: Pegylated Interferon and Ribavirin — Pegylated interefron is an injection and ribavirin is an oral tablet
  Other Names: Pegasys and Ribavirin
  Arms: 2

SUMMARY:
The GI-5005 therapeutic vaccine in combination with standard of care or standard of care alone will be injected under the skin of HCV subjects. Patients will be monitored for safety, immune responses and any therapeutic benefits related to the injections including EVR, ETR, and SVR.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection with genotype 1 based on serum positivity for HCV RNA or a positive test for serum anti-HCV antibody for at least 6 months;
* One of the following response criteria based on response to prior combination therapy with pegylated or non-pegylated interferon plus ribavirin:

Non-Responders

* Poor responders - a subset of non-responders who achieved > 1 log10 but < 2 log10 reduction in HCV RNA after a minimum of 12 weeks of prior interferon based therapy.
* Partial responders - a subset of non-responders who achieve at least a 2 log10 reduction in HCV RNA by 12 weeks, but do not achieve an end of treatment response (ETR defined as HCV RNA negativity by PCR assay at the end of a minimum of 6 months of therapy).

Naive

* Patients who are treatment naïve and have refused IFN therapy for reasons other than contraindication.
* Signed, written, informed consent from the patient or legal representative before any study-specific procedures are performed;
* Liver biopsy within 3 years of the screening visit, documenting extent of liver disease consistent with chronic hepatitis C with evidence of inflammation and/or fibrosis. Liver biopsy within 1 year for subjects consenting to paired biopsy testing. Eight unstained liver biopsy slides are required for the baseline sample and post-treatment sample for use in central blinded evaluation for paired biopsy testing;
* Age ≥ 18 years;
* Negative scratch test (immediate hypersensitivity, IgE mediated) to S. cerevisiae.

Exclusion Criteria:

* History of decompensated liver disease, including but not restricted to, portal hypertension as manifested by a known history of gastroesophageal varices, variceal bleeding, ascites or encephalopathy, histopathologic or clinical evidence of cirrhosis, hepatocellular carcinoma, or renal impairment consistent with hepatorenal syndrome;
* History of significant non-HCV chronic liver disease, i.e. alcoholic hepatitis, autoimmune hepatitis;
* Null response to prior IFN plus ribavirin therapy, defined as patients that have received at least 12 weeks of interferon-based treatment with < 1 log10 reduction in viral load;
* Subjects treated with more than 1 complete hepatitis C regimen (subjects with a history of 1 complete prior regimen and a second incomplete prior regimen may be eligible upon discussion with and approval of the medical monitor);
* Subjects that required a dose reduction of >25% of the planned exposure of IFN or >50% of their planned ribavirin exposure during their previous interferon/ribavirin treatment;
* Subjects that required growth factors during their previous interferon/ribavirin treatment;
* Subjects that received small molecule inhibitor therapy combined with an interferon based regimen. (subjects that received small molecule inhibitor monotherapy can be included);
* Treatment for HCV infection within 28 days before screening;
* Chronic hepatitis B infection or positive hepatitis B surface antigen (HBsAg) at screening;
* Body weight >275 pounds;
* Known history of HIV infection or positive HIV antibody test at screening;
* History of Crohn's disease or ulcerative colitis;
* Concurrent therapy with herbal supplements taken specifically for the treatment of HCV (i.e. milk thistle). Wash-out of HCV related herbals for 28 days prior to Day 1. Consult sponsor before excluding potential subjects;
* Alcohol and/or IV drug abuse within the past year;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Research and Education inc., San Diego, California
  - University of Colorado, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - University of Connecticut Health Center, Farmingtom, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - NW Georgia Research Institute, Marietta, Georgia
  - Hawaii Medical Center, Honolulu, Hawaii
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Tulane University Hospital, New Orleans, Louisiana
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Gastroenterology Associates, PA, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Liver Institute of Virginia Bon Secours Health System, Newport News, Virginia
  - McGuire VA Medical Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 Investigators in the U.S. (30 in U.S., 3 in Europe, 5 in India) were recruited to participate in this study. First subject was screened on November 12, 2007 and the last subject was screened on March 7, 2011.
Groups:
- Arm 1: Peg-IFN/Ribavirin Plus GI-5005: Subjects were given GI-5005 alone for 12 weeks (5 weekly followed by 2 monthly doses). After completion of GI-5005 monotherapy run in period peg-IFN/ribavirin (SOC) therapy was added to continued monthly administration of GI-5005 and the subjects were treated for subsequent 12 week period. At the end of this period, subjects who achieve an EVR continued to receive GI-5005 plus SOC therapy for an additional 36 weeks (naive subjects) or an additional 60 weeks (non-responder subjects). Subjects who did not achieve an EVR were followed for safety during a 36 week off treatment period. Any subject who discontinued SOC therapy due to intolerance at or prior to EVR assessment was treated with GI-5005 monotherapy for up to a total of 72 weeks.
- Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005: Subjects were treated with 12 weeks of SOC (Peg-IFN plus Ribavirin) therapy. Subjects who achieve an EVR continued to receive SOC therapy for an additional 36 weeks (naive subjects) or an additional 60 weeks (non-responder subjects). Subjects who did not achieve an EVR, GI-5005 was added to SOC therapy and study drug administration continued for up to an additional 62 weeks. Subjects who discontinued SOC therapy due to intolerance were treated with GI-5005 monotherapy for up to 72 weeks.
Period: Overall Study
Arm/Group | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005
Started | 72 | 68
Completed | 60 | 53
Not Completed | 12 | 15
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 4 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Non-compliance | 0 | 1
Not completed — Randomized, not treated | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005 | Total
Number analyzed (Participants) | 72 | 68 | 140
Age, Continuous [Median (Full Range); unit: years] | 48 [20 to 74] | 49 [20 to 68] | 48 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 42 | 45 | 87
Region of Enrollment [Number; unit: participants]
  United States | 62 | 62 | 124
  Europe | 6 | 4 | 10
  India | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: EVR (Early Virologic Response)
Description: Early Virologic Response (EVR) is a response measured by the reduction of virus in the blood after 12 weeks of treatment.
Time Frame: At 12 weeks of treatment
Population: One hundred forty subjects were randomized, only 133 subjects received at least one dose of study drug. Subjects who did not receive at least one dose of study drug were removed from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005
Number analyzed (Participants) | 68 | 65
percentage of participants | 79.4 | 78.5
Statistical Analysis 1: Comparison: Arm 1: Peg-IFN/Ribavirin Plus GI-5005 vs Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel test

ADVERSE EVENTS:
Arm/Group | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005
Serious Adverse Events (participants affected / at risk) | 14/71 | 7/65
Other Adverse Events (participants affected / at risk) | 70/71 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 (N=71) | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005 (N=65)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug abuser (Social circumstances) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Peg-IFN/Ribavirin Plus GI-5005 (N=71) | Arm 2: Peg-IFN/Ribavirin or Peg-IFN/Ribavirin Plus GI-5005 (N=65)
Anaemia (Blood and lymphatic system disorders) | 43 | 44
Leucopenia (Blood and lymphatic system disorders) | 4 | 3
neutropenia (Blood and lymphatic system disorders) | 57 | 51
Dry eye (Eye disorders) | 5 | 2
abdominal pain (Gastrointestinal disorders) | 10 | 8
abdominal pain upper (Gastrointestinal disorders) | 5 | 2
constipation (Gastrointestinal disorders) | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 15 | 18
Dry mouth (Gastrointestinal disorders) | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 7 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 6
Haemorrhoids (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 28 | 26
vomitting (Gastrointestinal disorders) | 14 | 9
Asthenia (General disorders) | 4 | 3
Chest pain (General disorders) | 5 | 5
Chills (General disorders) | 14 | 16
Fatigue (General disorders) | 44 | 46
Influenza like illness (General disorders) | 14 | 14
Injection site bruising (General disorders) | 6 | 1
Injection site erythema (General disorders) | 30 | 21
Injection site induration (General disorders) | 8 | 0
Injection site pain (General disorders) | 22 | 9
Injection site pruritus (General disorders) | 8 | 1
Injection site swelling (General disorders) | 7 | 1
Irritability (General disorders) | 16 | 18
Malaise (General disorders) | 6 | 1
Oedema peripheral (General disorders) | 5 | 4
Pain (General disorders) | 11 | 13
Pyrexia (General disorders) | 20 | 18
Hepatomegaly (Hepatobiliary disorders) | 1 | 5
Bronchitis (Infections and infestations) | 4 | 2
Herpes simplex (Infections and infestations) | 6 | 2
Nasopharyngitis (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 11 | 8
Urinary tract infection (Infections and infestations) | 9 | 6
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Excoriation (Injury, poisoning and procedural complications) | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 3
Neutrophil count decreased (Investigations) | 4 | 3
Weight decreased (Investigations) | 11 | 9
White blood cell count decreased (Investigations) | 4 | 2
anorexia (Metabolism and nutrition disorders) | 9 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Amnesia (Nervous system disorders) | 1 | 6
Disturbance in attention (Nervous system disorders) | 2 | 6
Dizziness (Nervous system disorders) | 10 | 14
Dysgeusia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 27 | 29
Hypoaesthesia (Nervous system disorders) | 0 | 4
Memory impairment (Nervous system disorders) | 7 | 0
Migraine (Nervous system disorders) | 6 | 0
Paraesthesia (Nervous system disorders) | 3 | 4
Anxiety (Psychiatric disorders) | 8 | 13
Depression (Psychiatric disorders) | 17 | 23
Insomnia (Psychiatric disorders) | 22 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 8
Dermititis (Skin and subcutaneous tissue disorders) | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6
Hypotrichosis (Skin and subcutaneous tissue disorders) | 1 | 5
Puritus (Skin and subcutaneous tissue disorders) | 12 | 15
Puritus generalized (Skin and subcutaneous tissue disorders) | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 19 | 16
Hypertension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will not publish or present in any forum any writing or discussion that involves Sponsor intellectual property or clinical trial information until the study has been finalized and all completed case report forms have been delivered to Sponsor. The confidentiality obligations will remain in effect for 5 years from the date of termination or expiration of study agreement.